CLINICAL TRIAL: NCT05742620
Title: Follow-up and Registration Study of Anlotinib Combined With Adjuvant Chemotherapy in the Treatment of Locally Advanced Gastrointestinal Tumors
Brief Title: Adjuvant Treatment of Digestive Tract Tumors
Acronym: ATDTT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQXB-GC-II-003
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Adjuvant Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib+CAPEOX/SOX (Experimental): Adjuvant treatment of locally advanced gastric cancer and colorectal cancer
  Interventions: Drug: anlotinib+CAPEOX/SOX

INTERVENTIONS:
Drug: anlotinib+CAPEOX/SOX — Patients with colorectal cancer use the anlotinib+CAPEOX protocol, and patients with gastric cancer use the anlotinib+SOX protocol.
  Anlotinib: 12mg, administered once a day on day 1-14, taken about half an hour before breakfast (the time of daily administration should be the same as much as possible), delivered with warm water, repeated once every three weeks;
  CAPEOX: capecitabine 1000mg/m2 each time, oral, twice a day, 1-14 days; Oxaliplatin: 130mg/m2 iv drip d1.
  SOX: Tegio: 100mg/day, continuous medication for 2 weeks, stop for 1 week; Oxaliplatin: 130mg/m2 iv drip d1.
  Other Names: anlotinib+chemotherapy

SUMMARY:
To evaluate the 3-year Disease-free survival rate(DFSR) of patients with locally advanced gastric cancer and colorectal cancer treated with anlotinib combined with adjuvant chemotherapy.

DETAILED DESCRIPTION:
Gastrointestinal tumor has a high incidence rate and mortality, which is one of the major diseases that seriously endanger the health of Chinese residents. Postoperative recurrence of colorectal cancer is the main cause of death in patients with advanced colorectal cancer. It is reported that the local recurrence rate after radical resection of colorectal cancer is 1% - 17%, and the 5-year survival rate after reoperation for recurrent and metastatic colorectal cancer is only 5% - 30%. In addition, the 5-year survival rate of locally advanced gastric cancer after operation is only 30-40%.

The adjuvant treatment of locally advanced colorectal cancer and gastric cancer is still mainly radiotherapy and chemotherapy, and the research of anti-vascular targeted therapy combined with adjuvant chemotherapy for locally advanced colorectal cancer and gastric cancer is still under exploration. The research of antiangiogenic drugs combined with adjuvant chemotherapy in the treatment of locally advanced colorectal cancer and gastric cancer can fill this gap. Therefore, this study was designed to explore the efficacy and safety of antiangiogenic drugs combined with adjuvant chemotherapy in the treatment of locally advanced colorectal cancer and gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.18 years old ≤ age ≤ 75 years old, male or female;
* 2. ECOG score 0~2 points;
* 3. Patients with locally advanced gastric cancer and colorectal cancer after radical surgery (R0 resection);
* 4. Gastric cancer: patients with stage III (pT1N3bM0, pT2N3M0, pT3N2-3M0, pT4aN1-3M0, pT4bN0-3M0);
* 5. Colorectal cancer: patients with stage III (T any N+M0);
* 6. Normal function of main organs
* 7. Female subjects of childbearing age must carry out a serum pregnancy test within 3 days before starting the study medication, and the result is negative, and are willing to use a medically approved effective contraceptive measure (such as intrauterine device, contraceptive or condom) during the study period and within 3 months after the last administration of the study medication; For male subjects whose partners are women of childbearing age, they should undergo surgical sterilization or agree to use effective methods of contraception during the study and within 3 months after the last study administration.
* 8. Subjects voluntarily joined the study and signed the informed consent form, with good compliance and cooperation in follow-up.

Exclusion Criteria:

* 1. Postoperative distal metastasis or failure to achieve R0 resection;
* 2. Have experienced any anti-tumor treatment before surgery, including chemotherapy, radiotherapy and targeted drug treatment;
* 3. Patients with contraindications to chemotherapy;
* 4. Other malignant tumors in the past 3 years;
* 5. Clinically obvious bleeding symptoms or obvious bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood++or above the baseline, or vasculitis);
* 6. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite the best drug treatment);
* 7. People newly diagnosed with angina pectoris within 3 months before screening or suffering from serious cardiovascular diseases within 6 months before screening, including unstable angina pectoris or myocardial infarction; Arrhythmias (including QTcF: male ≥ 450 ms, female ≥ 470 ms) require long-term use of antiarrhythmic drugs; ≥ Grade 2 congestive heart failure (NYHA classification);
* 8. Severe infection (such as the need for intravenous drip of antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first administration, or fever of unknown cause occurred during screening/before the first administration>38.5 ° C;
* 9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 10. Pregnant or lactating women; Those with fertility who are unwilling or unable to take effective contraceptive measures;
* 11. It is known that it will produce allergy, hypersensitivity or intolerance to the test drug and its excipients;
* 12. Subjects who are participating in other clinical studies or whose first medication is less than 4 weeks from the end of the previous clinical study (the last medication), or who have 5 half-lives of the study drug;
* 13. Subjects are known to have a history of abuse of psychotropic substances, alcohol or drug abuse;
* 14. The researcher believes that there are any conditions that may harm the subject or cause the subject to fail to meet or perform the research requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2029-07-20 (Estimated)

PRIMARY OUTCOMES:
3y-DFSR | 3years
  3-year Disease-free survival

SECONDARY OUTCOMES:
DFS | 3years
  Disease free survival
3y-OSR | 3years
  3-year Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: DeLiang Yu, Doctor, Study Chair — Ambulatory Surgery Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grothey A, Sobrero AF, Shields AF, Yoshino T, Paul J, Taieb J, Souglakos J, Shi Q, Kerr R, Labianca R, Meyerhardt JA, Vernerey D, Yamanaka T, Boukovinas I, Meyers JP, Renfro LA, Niedzwiecki D, Watanabe T, Torri V, Saunders M, Sargent DJ, Andre T, Iveson T. Duration of Adjuvant Chemotherapy for Stage III Colon Cancer. N Engl J Med. 2018 Mar 29;378(13):1177-1188. doi: 10.1056/NEJMoa1713709. PMID 29590544
- [Background] Andre T, Meyerhardt J, Iveson T, Sobrero A, Yoshino T, Souglakos I, Grothey A, Niedzwiecki D, Saunders M, Labianca R, Yamanaka T, Boukovinas I, Vernerey D, Meyers J, Harkin A, Torri V, Oki E, Georgoulias V, Taieb J, Shields A, Shi Q. Effect of duration of adjuvant chemotherapy for patients with stage III colon cancer (IDEA collaboration): final results from a prospective, pooled analysis of six randomised, phase 3 trials. Lancet Oncol. 2020 Dec;21(12):1620-1629. doi: 10.1016/S1470-2045(20)30527-1. PMID 33271092
- [Background] Petrelli F, Labianca R, Zaniboni A, Lonardi S, Galli F, Rulli E, Rosati G, Corallo S, Ronzoni M, Cardellino GG, Mattioli R, Mambrini A, Ciuffreda L, Banzi M, Pusceddu V, Maiello E, Zampino M, Zagonel V, Marchetti P, Corsi D, Rimassa L, Cinieri S, Sobrero A. Assessment of Duration and Effects of 3 vs 6 Months of Adjuvant Chemotherapy in High-Risk Stage II Colorectal Cancer: A Subgroup Analysis of the TOSCA Randomized Clinical Trial. JAMA Oncol. 2020 Apr 1;6(4):547-551. doi: 10.1001/jamaoncol.2019.6486. PMID 32053133
- [Background] Iveson TJ, Sobrero AF, Yoshino T, Souglakos I, Ou FS, Meyers JP, Shi Q, Grothey A, Saunders MP, Labianca R, Yamanaka T, Boukovinas I, Hollander NH, Galli F, Yamazaki K, Georgoulias V, Kerr R, Oki E, Lonardi S, Harkin A, Rosati G, Paul J. Duration of Adjuvant Doublet Chemotherapy (3 or 6 months) in Patients With High-Risk Stage II Colorectal Cancer. J Clin Oncol. 2021 Feb 20;39(6):631-641. doi: 10.1200/JCO.20.01330. Epub 2021 Jan 13. PMID 33439695
- [Background] Tanabe K, Fujii M, Nishikawa K, Kunisaki C, Tsuji A, Matsuhashi N, Takagane A, Ohno T, Kawase T, Kochi M, Yoshida K, Kakeji Y, Ichikawa W, Chin K, Terashima M, Takeuchi M, Nakajima T. Phase II/III study of second-line chemotherapy comparing irinotecan-alone with S-1 plus irinotecan in advanced gastric cancer refractory to first-line treatment with S-1 (JACCRO GC-05). Ann Oncol. 2015 Sep;26(9):1916-1922. doi: 10.1093/annonc/mdv265. Epub 2015 Jun 24. PMID 26109630